CLINICAL TRIAL: NCT04803643
Title: Investigation of Upper Extremity Exercise Capacity, Muscle Oxygenation, Balance and Physical Activity Level in Patients With Cystic Fibrosis
Brief Title: Upper Extremity Exercise Capacity, Muscle Oxygenation, Balance in Patients With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Meral Boşnak Güçlü, Prof. Dr., Gazi University
Other Study IDs: Gazi University 22
Record Dates: First submitted 2021-03-03; First posted 2021-03-18 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-04

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; upper extremity exercise capacity; muscle oxygenation; balance; physical activity
MeSH Terms: conditions — Cystic Fibrosis; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients: Upper extremity exercise capacity will be assessed using six minute pegboard ring test, functional exercise capacity using six minute walk test, muscle oxygenation using "Moxy" monitor, balance using "Biodex Balance System®" and Y balance test, physical activity using multi-sensor activity monitor, pulmonary function using spirometry, respiratory muscle strength using mouth pressure device, peripheral muscle strength using hand held dynamometer, respiratory muscle endurance using incremental threshold loading test, life quality using "The Revised Cystic Fibrosis Questionnaire (CFQ-R)" (Turkish version).
- Healthy controls: Upper extremity exercise capacity will be assessed using six minute pegboard ring test, functional exercise capacity using six minute walk test, muscle oxygenation using "Moxy" monitor, balance using "Biodex Balance System®" and Y balance test, physical activity using multi-sensor activity monitor, pulmonary function using spirometry, respiratory muscle strength using mouth pressure device, peripheral muscle strength using hand held dynamometer, respiratory muscle endurance using incremental threshold loading test, life quality using "The Revised Cystic Fibrosis Questionnaire (CFQ-R)" (Turkish version).

SUMMARY:
The primary aim of the study is to evaluate upper extremity exercise capacity, muscle oxygenation, balance and physical activity level in patients with cystic fibrosis.. The secondary aim of the study is assessment of functional exercise capacity, respiratory function, peripheral and respiratory muscle strength, respiratory muscle endurance, quality of life in patients with cystic fibrosis and compare them with healthy controls.

DETAILED DESCRIPTION:
Cystic fibrosis (CF) is an autosomal recessive genetic disease. Although it is a monogenetic type of disease, its phenotype varies widely. CF is characterized by progressive lung disease, malabsorption of fat and protein, fatty stools, pancreatic insufficiency resulting in gastrointestinal malabsorption, intestinal abnormalities resulting in malnutrition, growth retardation, sinusitis, and diabetes. The most important problems seen in patients are excessive secretion, decreased exercise capacity, dyspnea and muscle strength loss. Exercise capacity, respiratory functions, respiratory and peripheral muscle strength, respiratory muscle endurance, balance, physical activity, quality of life are poor in cystic fibrosis patients.There are insufficient studies on this subject in the literature. The number of studies using objective method is few. Cystic fibrosis patients have upper extremity muscle weakness. There is no study on the evaluation of upper extremity exercise capacity in these patients in the literature. Even if patients with CF have normal pulmonary function test results, there are studies showing that exercise intolerance has developed. These reasons have revealed the need to investigate oxygen metabolism at the cellular level.There are only two studies in the literature evaluating muscle oxygenation in patients with cystic fibrosis. There is no study evaluating with a "Moxy" monitor.The primary aim of the study is to evaluate upper extremity exercise capacity, muscle oxygenation, balance and physical activity level in patients with cystic fibrosis.. The secondary aim of the study is assessment of functional exercise capacity, respiratory function, peripheral and respiratory muscle strength, respiratory muscle endurance, quality of life in patients with cystic fibrosis and compare them with healthy controls.

The study was planned cross-sectional. At least 30 cystic fibrosis patients and 30 age- and sex-matched healthy controls will be included in the study. Individuals' exercise capacity, respiratory functions, physical activity levels, balance assessments, peripheral and respiratory muscle strength, respiratory muscle endurance, muscle oxygenation and quality of life will be evaluated. Upper extremity exercise capacity will be assessed using six minute pegboard ring test, functional exercise capacity using six minute walk test, muscle oxygenation using "Moxy" monitor, balance using "Biodex Balance System®" and Y balance test, physical activity using multi-sensor activity monitor, pulmonary function using spirometry, respiratory muscle strength using mouth pressure device, peripheral muscle strength using hand held dynamometer, respiratory muscle endurance using incremental threshold loading test, life quality using "The Revised Cystic Fibrosis Questionnaire (CFQ-R)" (Turkish version). The assessments will be completed in two days.

ELIGIBILITY:
Inclusion Criteria:

Patients;

* 6-18 years old
* Diagnosed with cystic fibrosis according to the American Cystic Fibrosis Association consensus report criteria
* Those who have not participated in the exercise training program planned in the last 3 months

Healthy controls;

* 6-18 years old

Exclusion Criteria:

Patients;

* A history of lung or liver transplant
* Diagnosed vision, hearing, vestibular, or neurological problems that can affect balance
* History of hospitalization previously (1 month)
* History of coronavirus disease (COVID-19)
* History of smoking
* Diagnosed orthopedic problems affecting mobility or a history of musculoskeletal surgery
* Acute pulmonary exacerbation
* Diagnosed with allergic
* Bronchopulmonary aspergillosis
* Systemic corticosteroids use
* Pulmonary hypertension and cardiovascular instability

Healthy controls;

* Trouble understanding and following the exercise test instruction
* A history of smoking

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: At least 30 patients with cystic fibroisis will be included in patients group and 30 healthy individuals will be included in control group
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Upper extremity exercise capacity | First Day
  Upper extremity exercise capacity will be evaluated with the 6-Minute Pegboard and Ring Test (Total number of rings). There are a total of 20 rings on the 4 iron bars on the board to be used. Patients will be asked to wear the rings with both hands first from top to bottom and then from bottom to top. At the end of 6 minutes, the total attached ring will be recorded in terms of pieces.

SECONDARY OUTCOMES:
Functional exercise capacity | First Day
  Functional exercise capacity will be evaluated with the 6- Minute Walk Test. 6- Minute Walk Test will be applied according to the American Thoracic Society (ATS) and European Respiratory Society (ERS) criteria.
Muscle Oxygenation | First Day
  Muscle oxygenation will be evaluated with the "Moxy" monitor (Moxy, Fortiori Design LLC, Minnesota, ABD). For measurement, "Moxy monitor" will be placed bilaterally at the 1/3 lower motor point of the quadriceps muscle group and on the deltoid muscle. A minimum of 3 minutes will be waited until the resting measurements and the skeletal muscle oxygenation (StO2) signal stabilize. The values (StO2 and total hemoglobin) will be recorded after the 6-minute walking test and the 6-Minute Pegboard and Ring Test. Data will be analyzed appropriately.
Balance | Second Day
  Static balance will be evaluated with the "Biodex Balance System®". Dynamic balance will be evaluated with the Y balance test. The data obtained from the system as a result of the test will be the general stability index, anterior / posterior (AP) stability index, medial / lateral (ML) stability index and their standard deviations. The tests will first be carried out on the hard ground with open eyes and then repeated on the soft ground. The measurements will then be repeated with eyes closed on hard and soft ground.
Physical activity (Total energy expenditure) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient will be informed about removing the device while taking a bath. Total energy expenditure (joule / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Active energy expenditure (joule / day)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient will be informed about removing the device while taking a bath. Active energy expenditure (joule / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Physical activity time (min / day)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient will be informed about removing the device while taking a bath. Physical activity time (min / day)will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Average metabolic equivalent (MET / day)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient will be informed about removing the device while taking a bath. Average metabolic equivalent (MET / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Number of steps (steps / day)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient will be informed about removing the device while taking a bath. Number of steps (steps / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Time spent lying down (min / day) days)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient will be informed about removing the device while taking a bath. Time spent lying down (min / day) days) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Physical activity (Sleep time (min / day)) | Second Day
  Physical activity will be evaluated with the Multi sensor activity monitor (SenseWear®, Inc Pittsburgh, ABD). The patient will wear the multisensor physical activity monitor over the triceps muscle of the non-dominant arm for 3 continuous days. The patient will be informed about removing the device while taking a bath. Sleep time (min / day) will be measured with the multi-sensor physical activity monitor. The parameters measured over two days will be averaged and analyzed with the "SenseWear® 7.0 Software" program.
Pulmonary function (Forced vital capacity (FVC)) | First Day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to ATS and ERS criteria. With the device, forced vital capacity (FVC) will be evaluated.
Pulmonary function (Forced expiratory volume in the first second (FEV1)) | First Day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to ATS and ERS criteria. With the device, forced expiratory volume in the first second (FEV1) will be evaluated.
Pulmonary function (FEV1 / FVC) | First Day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to ATS and ERS criteria. With the device, FEV1 / FVC will be evaluated.
Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) | First Day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to ATS and ERS criteria. With the device, flow rate 25-75% of forced expiratory volume (FEF 25-75%) will be evaluated.
Pulmonary function (Peak flow rate (PEF)) | First Day
  Pulmonary function will be evaluated with the spirometry. Dynamic lung volume measurements will be made according to ATS and ERS criteria. With the device, peak flow rate (PEF) will be evaluated.
Respiratory muscle strength | First Day
  Maximal inspiratory (MIP) and maximal expiratory (MEP) pressures expressing respiratory muscle strength will be measured with a portable mouth pressure measuring device according to ATS and ERS criteria.
Peripheral muscle strength | Second Day
  Isometric peripheral muscle strength will be measured with a portable hand dynamometer (JTECH Commander, USA). Measurements will be repeated on the shoulder abductors and knee extensors three times on the right and left.
Respiratory muscle endurance | Second Day
  Respiratory muscle endurance will be assessed by the POWERbreathe Wellness (POWERbreathe, Inspiratory Muscle Training (IMT) Technologies Ltd., Birmingham, UK) device and the respiratory muscle endurance test at increased threshold load. The test will be started with 20% of the maximal inspiratory pressure and the pressure will be increased to 40%, 60%, 80% and 100% every two minutes. Patients will be asked to continue breathing through the device during the test. During the test, the number of breaths delivered and the maximal time reached during each 2-minute period will be recorded. If the individual cannot breathe 3 consecutive times, the test will be terminated by the physiotherapist. The total duration of the test and the maximum pressure value at which it continues to breathe for at least 1 minute will be multiplied. The value found will be recorded as the respiratory muscle endurance value.
Life quality | Second Day
  Quality of life will be evaluated with the Turkish adaptation of the Revised Cystic Fibrosis Questionnaire (CFQ-R). The scale have well-established reliability and validity. There are four CFQ-R questionnaires for patients of three different age groups (6-10, 12-13, and 14 years and older). The CFQ-R children's version consists of 35 questions. Scale subtitles; It consists of physical functioning, emotional functioning, social functioning, body ımage, eating disorders, treatment burden, and respiratory and digestive symptoms. Items for child CFQ-R are rated according to a 4-point scale. Higher scores indicate better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Betül YOLERİ, Pt, Study Chair — Gazi University; Meral BOŞNAK GÜÇLÜ, Prof.Dr., Study Director — Gazi University; Ayşe TANA ARSLAN, Prof.Dr., Principal Investigator — Gazi University; Tuğba ŞİŞMANLAR EYÜBOĞLU, Asc. Prof.Dr, Principal Investigator — Gazi University
Locations (2):
- Turkey (Türkiye) (2):
  - Gazi University Faculty of Health Science Department of Physiotherapy and Rehabilitation, Ankara
  - Gazi University Faculty of Health Sciences Department of Physical Therapy and Rehabilitation, Ankara, Çankaya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sharma R, Florea VG, Bolger AP, Doehner W, Florea ND, Coats AJ, Hodson ME, Anker SD, Henein MY. Wasting as an independent predictor of mortality in patients with cystic fibrosis. Thorax. 2001 Oct;56(10):746-50. doi: 10.1136/thorax.56.10.746. PMID 11562511
- [Background] Arikan H, Yatar I, Calik-Kutukcu E, Aribas Z, Saglam M, Vardar-Yagli N, Savci S, Inal-Ince D, Ozcelik U, Kiper N. A comparison of respiratory and peripheral muscle strength, functional exercise capacity, activities of daily living and physical fitness in patients with cystic fibrosis and healthy subjects. Res Dev Disabil. 2015 Oct-Nov;45-46:147-56. doi: 10.1016/j.ridd.2015.07.020. Epub 2015 Aug 1. PMID 26241869
- [Background] Erickson ML, Seigler N, McKie KT, McCully KK, Harris RA. Skeletal muscle oxidative capacity in patients with cystic fibrosis. Exp Physiol. 2015 Apr 20;100(5):545-52. doi: 10.1113/EP085037. PMID 25758606
- [Background] Schneiderman JE, Wilkes DL, Atenafu EG, Nguyen T, Wells GD, Alarie N, Tullis E, Lands LC, Coates AL, Corey M, Ratjen F. Longitudinal relationship between physical activity and lung health in patients with cystic fibrosis. Eur Respir J. 2014 Mar;43(3):817-23. doi: 10.1183/09031936.00055513. Epub 2013 Oct 31. PMID 24176992
- [Background] Santana NN, Chaves CRMM, Goncalves CP, Gomes Junior SCDS. FACTORS ASSOCIATED TO QUALITY OF LIFE IN CHILDREN AND ADOLESCENTS WITH CYSTIC FIBROSIS. Rev Paul Pediatr. 2020 Jun 19;38:e2018397. doi: 10.1590/1984-0462/2020/38/2018397. eCollection 2020. PMID 32578674